CLINICAL TRIAL: NCT00750737
Title: Phase III Clinical Trial of Oral Posaconazole 3 Times/Day vs Weekly High Dose Amphotericin B Lipid Complex (ABLC) for Prevention of Invasive Fungal Infections In Patients With Hematologic Malignancies & Hematopoietic Stem Cell Transplant
Brief Title: Oral Posaconazole Three Times Per Day vs Weekly High Dose Amphotericin B Lipid Complex (ABLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Enzon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0020
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Results first posted 2016-01-06 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-01

CONDITIONS: Invasive Fungal Infections; Hematologic Malignancies
Keywords: Hematologic Malignancies; Blood Cancer; Lymphatic Cancer; Amphotericin B Lipid Complex; Amphotericin B; ABLC; Fungizone; Noxafil; SCH56592; Posaconazole; Invasive fungal infections; IFI; Hematopoietic Stem Cell Transplant; HSCT; Bone Marrow Transplant; Allogeneic hematopoietic stem cell transplant
MeSH Terms: conditions — Invasive Fungal Infections; Hematologic Neoplasms | interventions — posaconazole; Amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Posaconazole (Experimental): Posaconazole 200 mg three times daily by mouth up to 6 weeks (Days 1-42)
  Interventions: Drug: Posaconazole
- Amphotericin B Lipid Complex (ABLC) (Experimental): 7.5 mg/kg of ABLC intravenously infused over 4-6 hours once per week, for up to 6 weeks (from Day 1 through Day 42)
  Interventions: Drug: ABLC

INTERVENTIONS:
Drug: Posaconazole — 200 mg three times daily by mouth up to 6 weeks (Days 1-42)
  Other Names: SCH56592; Noxafil
  Arms: Posaconazole
Drug: ABLC — 7.5 mg/kg of ABLC intravenously infused over 4-6 hours once per week, for up to 6 weeks (from Day 1 through Day 42)
  Other Names: Amphotericin B Liquid Complex; Fungizone
  Arms: Amphotericin B Lipid Complex (ABLC)

SUMMARY:
The objective of this study is to compare the safety and efficacy of ABLC versus oral Posaconazole in the prevention of invasive fungal infections in high risk patients with hematologic malignancies or hematopoietic stem cell transplant.

Primary objective is to demonstrate the low toxicity rate and low rate of invasive fungal infections associated with ABLC or Posaconazole prophylaxis.

Secondary objective will be to compare the cost effectiveness of these two prophylactic regimens.

DETAILED DESCRIPTION:
The Study Drugs:

ABLC is an antifungal drug that is commonly used to treat and/or prevent a variety of serious invasive fungal infections (IFIs). In this study, ABLC will be used for IFI prevention.

Posaconazole is a newer antifungal drug that is commonly used to prevent serious IFIs.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to receive either posaconazole or ABLC. You will have an equal chance (50/50) of being assigned to either group. You and your study doctor will know which group you are in.

Study Drug Administration:

If you are assigned to the Posaconazole Group, you will take posaconazole 3 times a day by mouth for up to 6 weeks (Days 1-42). The study doctor will advise you about taking it with fatty meals and/or nutritional supplements.

If you are assigned to the ABLC Group, you will receive ABLC once a week by vein over 4-6 hours, for up to 6 weeks (from Day 1 through Day 42). If the creatinine level increases, the dose will be divided into 2 doses per week. The drug may be given in the hospital (if you are admitted to the hospital before or during the study) or at an outpatient treatment center.

Study Visits:

Once a week from Day 1 to Day 42, you will have the following procedures performed:

* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will be asked about any medications and treatments you may be receiving.
* You will be asked about any IFI symptoms that may have developed. You will also be asked about any side effects that may have occurred since your last visit. (You should contact the study doctor and/or study staff right away, if at any time you feel you have had a side effect.)

You may have certain routine diagnostic tests performed at any time in the study, if necessary to confirm you do not have an IFI. These tests may include blood collection (about 1 tablespoon), scans, skin tissue biopsy, and/or bronchoscopy.

Length of Study:

You will receive study treatment for up to 6 weeks (42 days). If you develop an IFI or any intolerable side effects, you will be taken off study early. You may also be taken off study if your neutrophil (a type of white blood cell) counts recover.

End-of-Treatment Visit:

Your End-of-Treatment visit will be on the last day you received the study drug (at most, 42 days after you started). The following procedures will be performed.

* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will have a physical exam, including measurement of vital signs.
* If the study doctor and/or your primary doctor thinks you may have an IFI, routine diagnostic tests may be performed.

Follow-up Visit:

Your follow up visit will be completed 7 - 14 days after your end-of-treatment visit. The following procedures will be performed:

* You will be checked for any signs of IFI.
* If your doctor suspects you have an IFI, a scan (such as an x-ray or CT scan) and/or bronchoscopy may be performed.
* You will be asked about any medications and treatments you may be receiving, and any side effects you may have had.
* Your vital signs will be checked, and a physical exam may be performed.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* An ECG may be performed.

This is an investigational study. ABLC and posaconazole are FDA approved and commercially available for the treatment and prevention of IFIs. Posaconazole is FDA approved for the way it is being used in this study. The study dose and study schedule for ABLC, however, is considered experimental. Currently, this dose and schedule for ABLC is being used in research only.

Up to 100 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects: 18 years of age or above.
2. Any allogeneic hematopoietic stem cell transplant (HSCT) patient who is at risk of invasive fungal infection (IFI) within 6 months of the transplant will be eligible for the study according to HSCT institutional anti-fungal prophylaxis guidelines.
3. Subjects must be willing to give written informed consent and able to adhere to dosing and study visit schedule.
4. Female subjects of childbearing potential must have a negative serum pregnancy test (beta-human chorionic gonadotropin [hCG]) at Baseline or within 96 hours before the start of study drug.
5. Female subjects of childbearing potential must agree to use a medically accepted method of contraception prior to screening, while receiving protocol-specified medication, and for 30 days after stopping the medication. Acceptable methods of contraception include condoms with/without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed IUD (intrauterine device), oral/injectable hormonal contraceptive, surgical sterilization (e.g. hysterectomy/tubal ligation).

Exclusion Criteria:

1. Subjects previously treated with antifungal therapy (voriconazole, fluconazole, or itraconazole) for proven or probable IFI within 30 days of enrollment.
2. Subjects who have taken the following drugs: terfenadine, cisapride, primazide, and ebastine; that are known to interact with azoles and that may lead to life-threatening side effects, within 24 hours before study drug administration. And astemizole within 7 days before study drug administration.
3. Subjects who have taken the following drugs: cimetidine, rifampin, carbamezapine, phenytoin, rifabutin, barbiturates, isoniazid, and vinca alkaloids (vincristine, vinblastine); that are known to lower the serum concentration/efficacy of azole antifungal agents, within 24 hours before study drug administration.
4. Subjects with a history of hypersensitivity or idiosyncratic reactions to azole agents or Amphotericin B.
5. Subjects on other nephrotoxic agents (e.g. foscarnet).
6. Patients who are unable to take pills.
7. Subjects with proven or probable invasive fungal infection.
8. Subjects with renal insufficiency (estimated creatine clearance less than 50mL/minute at Baseline or likely to require dialysis during the study).
9. Subjects having ECG with a prolonged QTc interval by manual reading: QTc greater than 500 msec. at Baseline.
10. Subjects with moderate or severe liver dysfunction at baseline, defined as aspartate amniotransferase (AST), alanine amniotransferase (ALT) and / or a total bilirubin level greater than 3 times the upper limit of normal (ULN).
11. Women who are breast feeding, pregnant, or intend to become pregnant during the course of the study.
12. Prior enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issam Raad, MD/Professor, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chaftari AM, Hachem RY, Ramos E, Kassis C, Campo M, Jiang Y, Prince RA, Wang W, Raad II. Comparison of posaconazole versus weekly amphotericin B lipid complex for the prevention of invasive fungal infections in hematopoietic stem-cell transplantation. Transplantation. 2012 Aug 15;94(3):302-8. doi: 10.1097/TP.0b013e3182577485. PMID 22814329
- See also: The University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 2008 to May 2009. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: A total of 46 participants were randomized, out of which 40 participants were included in the analysis and 6 participants withdrew consent.
Groups:
- Posaconazole 200 mg Oral: Posaconazole 200 mg three times daily by mouth up to 6 weeks (Days 1-42)
- Amphotericin B Lipid Complex (ABLC) 7.5 mg/kg IV: 7.5 mg/kg of ABLC intravenously infused over 4-6 hours once per week, for up to 6 weeks (from Day 1 through Day 42)
Period: Overall Study
Arm/Group | Posaconazole 200 mg Oral | Amphotericin B Lipid Complex (ABLC) 7.5 mg/kg IV
Started | 24 | 22
Completed | 21 | 19
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Posaconazole 200 mg Oral | Amphotericin B Lipid Complex (ABLC) 7.5 mg/kg IV | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Continuous [Median (Full Range); unit: years] | 55.5 [21 to 67] | 56 [22 to 70] | 55.5 [21 to 70]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 20 | 43
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 18
  Male | 19 | 9 | 28
Region of Enrollment [Number; unit: participants]
  United States | 24 | 22 | 46

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Invasive Fungal Infection (IFI)
Description: Percentage of participants that developed IFI within 7 days of antifungal prophylaxis therapy (Posaconazole or ABLC).
Time Frame: Within 7 days of antifungal prophylaxis therapy
Population: Out of 46 participants, 40 were included in the analysis and 6 withdrew consent.
Measure: Number; unit: percentage of participants
Arm/Group | Posaconazole 200 mg Oral | Amphotericin B Lipid Complex (ABLC) 7.5 mg/kg IV
Number analyzed (Participants) | 21 | 19
percentage of participants | 0 | 5

2. Secondary Outcome: Efficacy Outcome Measured as Success or Failure
Description: Success: Defined as the absence of proven or probable invasive fungal infection through the end of prophylaxis and absence of Grade 1-4 toxicity related to prophylaxis requiring the discontinuation of the drug. Failure: Presence of proven or probable fungal infection or development of Grade 1-4 toxicity related to prophylaxis while on study drug and requiring discontinuation of study drug or inability to tolerate intravenous ABLC (due to infusion related toxicities) or oral Posaconazole (due to mucositis or vomiting).
Time Frame: Day 1 through Day 42
Population: Out of 46 participants, 40 were included in the analysis and 6 withdrew consent.
Measure: Number; unit: percentage of participants
Arm/Group | Posaconazole 200 mg Oral | Amphotericin B Lipid Complex (ABLC) 7.5 mg/kg IV
Number analyzed (Participants) | 21 | 19
percentage of participants
  Success | 62 | 21
  Failure | 38 | 79

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were evaluated from the time of the first infusion of study drug through the end of the post-treatment visit. Collection period: July 10, 2008 to July 31, 2009.
Arm/Group | Posaconazole 200 mg Oral | Amphotericin B Lipid Complex (ABLC) 7.5 mg/kg IV
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 21/21 | 19/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole 200 mg Oral (N=21) | Amphotericin B Lipid Complex (ABLC) 7.5 mg/kg IV (N=19)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (6) | 8 (8)
Chills (General disorders) | 1 (1) | 6 (6)
Increase in ALT (Metabolism and nutrition disorders) | 10 (10) | 5 (5)
Increase in Bilirubin (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
Nausea (Gastrointestinal disorders) | 14 (14) | 10 (10)
Vomiting (Gastrointestinal disorders) | 6 (6) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 14 (14) | 8 (8)
Invasive Fungal Infection (Infections and infestations) | 0 (0) | 1 (1)
Increase in Creatinine (Metabolism and nutrition disorders) | 5 (5) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No